CLINICAL TRIAL: NCT02257606
Title: Robot-assisted Training on the Upper Limb in Persons With MS: an RCT
Brief Title: Robot-assisted Training of the Upper Limb in Persons With Multiple Sclerosis: an Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); Expertise Centre for digital Media (Unknown); tUL (Unknown); iMinds (Industry); Interreg (Other)
Responsible Party: Principal Investigator, Peter Feys, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CME2011/315
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (persons with MS) (No Intervention): no training
- Experimental group (persons with MS) (Experimental): Robot-assisted training
  Interventions: Other: I-TRAVLE training

INTERVENTIONS:
Other: I-TRAVLE training
  Arms: Experimental group (persons with MS)

SUMMARY:
With this randomised intervention study, the investigators want to investigate the training effect of an 8 week training regime, using a robot-assisted training system in persons with MS. Besides conventional therapy, study participants in the experimental group will train 3 times per week during 30 minutes, using the haptic master. Research questions focus on the effects of additional robot assisted training on range of motion, movement quality and clinical tests for the upper limb in persons with MS. Evaluation by means of questionnaires and clinical outcome measures occured at baseline, after 4 weeks, after 8 weeks and at 16 weeks of follow-

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Multiple Sclerosis (McDonald criteria), upper limb dysfunction due to muscle weakness (Motricity Index <80), age > 18 years

Exclusion Criteria:

* MS relapse or glucocorticosteroid treatment in the last month before the start of the study, upper limb paralysis (Motricity Index < 18), other sever limitations, influencing participation (cognitive, visual)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Motricity index | 2.5 min (pre-post)
  Random motor activity
Fugl-Meyer | 30 min (pre-post)
  Assessment of recovery of motor function
Action Research arm test | 15-20 min (pre-post)
  Grasp, grip, pinch, gross movement
Motor Activity log | 45 min (pre-post)
  perceived activities of daily life
Jamar handgrip strength | 2.5 min (pre-post)
  Handgrip strength

REFERENCES:
- [Derived] Feys P, Coninx K, Kerkhofs L, De Weyer T, Truyens V, Maris A, Lamers I. Robot-supported upper limb training in a virtual learning environment : a pilot randomized controlled trial in persons with MS. J Neuroeng Rehabil. 2015 Jul 23;12:60. doi: 10.1186/s12984-015-0043-3. PMID 26202325